CLINICAL TRIAL: NCT02609984
Title: A Randomized, Open-Label, Phase 2 Trial of CMB305 (Sequentially Administered LV305 and G305) and Atezolizumab in Patients With Locally Advanced, Relapsed, or Metastatic Sarcoma Expressing NY-ESO-1
Brief Title: Study to Compare the Safety and Efficacy of CMB305 With Atezolizumab to Atezolizumab Alone in Participants With Sarcoma (IMDZ-C232/V943A-002)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study did not meet the efficacy objective
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMDZ-C232; V943A-002 (Other: Merck); IMDZ-C232 (Other: Immune Design)
Record Dates: First submitted 2015-11-14; First posted 2015-11-20 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma; Myxoid/Round Cell Liposarcoma; Synovial Sarcoma; Metastatic Sarcoma; Recurrent Adult Soft Tissue Sarcoma; Locally Advanced Sarcoma; Liposarcoma
Keywords: immunotherapy; CMB305; LV305; GLA-SE; atezolizumab; NY-ESO-1
MeSH Terms: conditions — Sarcoma; Liposarcoma, Myxoid; Sarcoma, Synovial; Liposarcoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CMB305 (sequentially administered LV305 and G305)+Atezolizumab (Experimental): Participants received CMB305 treatment in combination with 1200 mg/day atezolizumab administered by intravenous (IV) infusion every 3 weeks (Q3W) for up to approximately 2 years. CMB305 treatment consisted of 2 doses of LV305 administered intradermally (ID) on Days 0 and 14 followed every 2 weeks with alternating doses of G305 administered intramuscularly (IM) and LV305. LV305 was administered at a dose of 1×10^10 vector genomes and G305 at a dose of 5 mcg glucopyranosyl lipid A stable emulsion mixed with 250 mcg of NY ESO-1 protein.
  Interventions: Biological: CMB305; Biological: atezolizumab
- Atezolizumab (Active Comparator): Participants received 1200 mg/day atezolizumab by IV infusion Q3W for up to approximately 2 years.
  Interventions: Biological: atezolizumab

INTERVENTIONS:
Biological: CMB305 — A combination of LV305 administered intradermally (ID) and G305 administered intramuscularly (IM)
  Arms: CMB305 (sequentially administered LV305 and G305)+Atezolizumab
Biological: atezolizumab — IV Infusion
  Other Names: TECENTRIQ®

SUMMARY:
This is an open-label Phase 2 randomized study that will examine the use of the study agents, CMB305 (sequentially administered LV305 which is a dendritic cell-targeting viral vector expressing the New York Esophageal Squamous Cell Carcinoma 1 gene [NY-ESO-1] and G305 which is a NY-ESO-1 recombinant protein plus glucopyranosyl lipid adjuvant-stable emulsion [GLA-SE]) in combination with atezolizumab or atezolizumab alone, in participants with locally advanced, relapsed or metastatic sarcoma (synovial or myxoid/round cell liposarcoma) expressing the NY-ESO-1 protein.

There is no formal primary hypothesis for this study.

DETAILED DESCRIPTION:
This study is designed to investigate and examine the time to progression and overall survival for CMB305 in combination with atezolizumab or atezolizumab alone in the treatment of participants with sarcoma expressing NY-ESO-1 protein.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, relapsed, or metastatic sarcoma with measurable tumor burden following therapy, as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1); the total of all lesions must be ≤12 cm (for synovial sarcoma) or ≤15 cm (for myxoid/round cell liposarcoma [MRCL])
* Tumor histology consistent with synovial sarcoma or MRCL
* Tumor specimen positive for NY-ESO-1 expression by immunohistochemistry (IHC)
* Inadequate response, relapse, and/or unacceptable toxicity with ≥1 prior systemic, surgical, or radiation cancer therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Investigational therapy within 4 weeks prior to CMB305 dosing
* Prior administration of other NY-ESO-1-targeting immunotherapeutics
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), anti-programmed cell death receptor 1 (PD-1), and anti-programmed cell death ligand (PD-L1) therapeutic antibodies, or any other antibody or drug targeting T-cell costimulation
* Treatment with systemic immunostimulatory agents (including but not limited to interleukin-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to first dose
* Significant immunosuppression
* Other cancer therapies, including chemotherapy, radiation, biologics or kinase inhibitors within 3 weeks prior to the first scheduled dosing
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), risk of pulmonary toxicity, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* History of other cancer within 3 years
* Evidence of active tuberculosis or recent (<1 week prior to first scheduled dosing) clinically significant infection requiring systemic therapy
* Evidence of active hepatitis B (HepB), hepatitis C (HepC), or Human Immunodeficiency Virus (HIV) infection
* Known active or untreated central nervous system (CNS) metastases
* Pregnant, planning to become pregnant within 6 months of treatment, or nursing
* Known allergy(ies) to any component of CMB305, atezolizumab, or severe allergic reactions to monoclonal antibodies, fusion proteins, or Chinese hamster ovary (CHO) cell products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-04-29 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Stanford University Medical Center, Palo Alto, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic of Jacksonville, Jacksonville, Florida
  - Georgia Cancer Specialists, Sandy Springs, Georgia
  - Northwestern University Feinburg School of Medicine, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Monter Cancer Research, Lake Success, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Fox Chase cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Vermont Cancer Center, Burlington, Vermont
  - Scca/Fhcrc, Seattle, Washington

REFERENCES:
- [Derived] Chawla SP, Van Tine BA, Pollack SM, Ganjoo KN, Elias AD, Riedel RF, Attia S, Choy E, Okuno SH, Agulnik M, von Mehren M, Livingston MB, Keedy VL, Verschraegen CF, Philip T, Bohac GC, Yurasov S, Yakovich A, Lu H, Chen M, Maki RG. Phase II Randomized Study of CMB305 and Atezolizumab Compared With Atezolizumab Alone in Soft-Tissue Sarcomas Expressing NY-ESO-1. J Clin Oncol. 2022 Apr 20;40(12):1291-1300. doi: 10.1200/JCO.20.03452. Epub 2021 Jul 14. PMID 34260265

RESULTS

PARTICIPANT FLOW:
Groups:
- CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab: Participants received CMB305 treatment in combination with 1200 mg/day atezolizumab administered by intravenous (IV) infusion every 3 weeks (Q3W) for up to approximately 2 years. CMB305 treatment consisted of 2 doses of LV305 administered intradermally (ID) on Days 0 and 14 followed every 2 weeks with alternating doses of G305 administered intramuscularly (IM) and LV305. LV305 was administered at a dose of 1×10^10 vector genomes and G305 at a dose of 5 mcg glucopyranosyl lipid A stable emulsion mixed with 250 mcg of New York Esophageal Squamous Cell Carcinoma 1 (NY ESO-1) protein.
Period: Overall Study
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Started | 45 | 44
Treated | 45 | 43
Completed | 1 | 5
Not Completed | 44 | 39
Not completed — Death | 29 | 26
Not completed — Participation Discontinued by Sponsor | 12 | 10
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disease Progression | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab: Participants received CMB305 treatment in combination with 1200 mg/day atezolizumab administered by IV infusion Q3W for up to approximately 2 years. CMB305 treatment consisted of 2 doses of LV305 administered ID on Days 0 and 14 followed every 2 weeks with alternating doses of G305 administered IM and LV305. LV305 was administered at a dose of 1×10^10 vector genomes and G305 at a dose of 5 mcg glucopyranosyl lipid A stable emulsion mixed with 250 mcg of NY ESO-1 protein.
- Total: Total of all reporting groups
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (16.52) | 46.7 (14.06) | 46.4 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 37 | 34 | 71
  Unknown or Not Reported | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The race is presented for all participants.
  Participants
    Race: White | 35 | 38 | 73
    Race: Asian | 3 | 1 | 4
    Race: Black or African American | 1 | 3 | 4
    Race: American Indian or Alaska Native | 2 | 0 | 2
    Race: Native Hawaiian or Other | 2 | 0 | 2
    Race: Other | 2 | 0 | 2
    Race: Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first, per RECIST 1.1 modified to use immune-related response criteria (irRC) confirmation and unidimensional tumor measurements as assessed by Blinded Independent Central Review (BICR). PD was defined as ≥20% increase in tumor burden compared with nadir (at any single time point) in 2 consecutive observations ≥4 weeks apart. If there was no disease progression or death, participants were censored at the date of their last disease assessment. The PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 36.1 months
Population: The analysis population included all randomized participants who met eligibility criteria for the study and had data recorded in the electronic Case Report Form (eCRF). Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Months | 2.6 [1.4 to 2.9] | 1.6 [1.5 to 2.7]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.4900, Log Rank — P-value based on a 2-sided stratified log-rank test stratified by type of sarcoma: synovial sarcoma versus myxoid/round cell liposarcoma; Hazard Ratio (HR) = 0.8568, 95% CI 2-sided [0.5507 to 1.3330] — Hazard ratio is from Cox proportional hazards model stratified by type of sarcoma: synovial sarcoma versus myxoid/round cell liposarcoma

2. Primary Outcome: Overall Survival (OS)
Description: OS was determined for all participants and was defined as the time from randomization to death due to any cause. Participants were censored at the date of their last follow-up. The OS was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 36.1 months
Population: The analysis population included all randomized participants who met eligibility criteria for the study and had data recorded in the eCRF. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Months | 18.2 [10.1 to 22.1] | 18.0 [15.3 to 26.5]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.4737, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.2145, 95% CI 2-sided [0.7131 to 2.0684] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Experiencing a Dose-Limiting Toxicity (DLT)
Description: DLTs will be evaluated during the safety run-in period. Any treatment emergent Grade 3 or higher adverse event (AE) that occurs in the first 42 days after initiation of study treatment, that is deemed possibly, probably or definitely related to the combination of CMB305 and atezolizumab will be considered a DLT with the following exceptions:
  * Alopecia or vomiting (unless not controlled by optimal anti-emetics)
  * Hepatic enzyme elevations associated with the baseline Grade 2 abnormalities
  * Grade 3 laboratory AEs that are asymptomatic and return to baseline or to Grade 1 within 3 days, unless identified specifically as DLT by the investigator or the Data Monitoring Committee (DMC)
  * Grade 3 fatigue
  * Grade 3 systemic reactions (such as fever, headache, influenza like symptoms, myalgia, malaise, or nausea) that return to baseline or Grade 1 within 3 days of study inoculation
Time Frame: Up to approximately 42 days
Population: The analysis population included all participants who participated in the safety run-in period and received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

4. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 36.1 months
Population: The analysis population included all participants who received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 43
Participants | 44 | 43

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 43
Participants | 6 | 6

6. Secondary Outcome: Progression-Free Survival (PFS) Rate at Month 3 Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first, per RECIST 1.1 modified to use irRC confirmation and unidimensional tumor measurements as assessed by BICR. PD was defined as ≥20% increase in tumor burden compared with nadir (at any single time point) in 2 consecutive observations ≥4 weeks apart. If there was no disease progression or death, participants were censored at the date of their last disease assessment. The PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data. Participants were evaluated every 6 weeks with radiographic imaging to assess their response to treatment. The PFS rate was calculated as the percentage of participants with PFS at Month 3.
Time Frame: Month 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Percentage of participants | 32.6 [19.4 to 46.4] | 23.8 [12.4 to 37.4]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.3645, Log Rank — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Progression-Free Survival (PFS) Rate at Month 6 Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first, per RECIST 1.1 modified to use irRC confirmation and unidimensional tumor measurements as assessed by BICR. PD was defined as ≥20% increase in tumor burden compared with nadir (at any single time point) in 2 consecutive observations ≥4 weeks apart. If there was no disease progression or death, participants were censored at the date of their last disease assessment. The PFS was analyzed using the product-limit (Kaplan-Meier) method for censored data. Participants were evaluated every 6 weeks with radiographic imaging to assess their response to treatment. The PFS rate was calculated as the percentage of participants with PFS at Month 6.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Percentage of participants | 16.5 [7.0 to 29.6] | 9.5 [3.0 to 20.6]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.3466, Log Rank — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to Next Treatment (TTNT)
Description: TTNT was the time from date of randomization to the start date of subsequent treatment. Participants were treated for up to approximately 2 years and then followed until next treatment or death. Participants who did not receive subsequent treatment were censored at the date of last contact or death. The TTNT was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 36.1 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 43
Months | 6.2 [4.4 to 9.1] | 4.9 [3.3 to 6.4]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.1622, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.7006, 95% CI 2-sided [0.4241 to 1.1574] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Distant Metastasis Free Survival (DMFS)
Description: DMFS was the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first. Participants without metastasis and death were censored at the date of last contact or death. The DMFS was analyzed using the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to approximately 36.1 months
Population: as for outcome 2
Measure: Median (Full Range); unit: Months
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Months | 5.3 [0.0 to 23.5] | 5.5 [0.0 to 31.8]
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.6397, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.1849, 95% CI 2-sided [0.5817 to 2.4134] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants Positive for Anti-New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) Antibody at Baseline
Description: The number of participants with anti-NY-ESO-1 antibodies at baseline was measured using an enzyme-linked immunosorbent assay (ELISA) with recombinant NY-ESO1 protein. A titer of >1:100 was considered positive. The number of participants that were anti-NY-ESO-1 antibody positive at baseline is presented.
Time Frame: Baseline (Day 1)
Population: The analysis population included all participants who received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab and had data available for baseline antibody analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 35 | 29
Participants | 14 | 6
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.1128, exact Pearson chi-square test

11. Secondary Outcome: Number of Participants Positive for Anti-New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) Antibody After Induction With Treatment
Description: The number of participants with anti-NY-ESO-1 antibodies induced after treatment was measured using an enzyme-linked immunosorbent assay (ELISA) with recombinant NY-ESO1protein. A titer of >1:100 was considered positive. The induction of anti-NY-ESO-1 antibody response was deﬁned as a ≥4-fold increase in the titer or the presence of a newly positive response after the ﬁrst dose of treatment. The number of participants that were anti-NY-ESO-1 antibody positive after induction with treatment is presented.
Time Frame: Up to approximately 24 months
Population: The analysis population included all participants who received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab and had data available for induction after treatment antibody analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 32 | 27
Participants | 16 | 0
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p < 0.0001, exact Pearson chi-square test

12. Secondary Outcome: Number of Participants Positive for Anti-New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) T Cells at Baseline
Description: Anti-NY-ESO-1 CD4 and CD8 positive T-cell responses were measured by interferon gamma detecting enzyme-linked ImmunoSpot (ELISPOT) using isolated CD4 and CD8 positive T cells from peripheral blood mononuclear cells (PBMCs) expanded in vitro with a NY-ESO-1 peptide pool (20-mer peptides, 10-mer overlap) and considered positive if there were >50 spot-forming units/50,000 cells observed for NY-ESO-1 peptides and a ≥2-fold increase in spot-forming units compared with a negative control. The number of participants that were anti-NY-ESO-1 T cell positive at baseline is presented.
Time Frame: Baseline (Day 1)
Population: The analysis population included all participants who received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab and had data available for baseline T cell analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 27 | 24
Participants | 17 | 12
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.4050, exact Pearson chi-square test

13. Secondary Outcome: Number of Participants Positive for Anti-New York Esophageal Squamous Cell Carcinoma-1 (NY-ESO-1) T Cells After Induction With Treatment
Description: Anti-NY-ESO-1 CD4 and CD8 positive T-cell responses were measured by interferon gamma detecting enzyme-linked ImmunoSpot (ELISPOT) using isolated CD4 and CD8 positive T cells expanded with a NY-ESO-1 peptide (20-mer peptides, 10-mer overlap) and considered positive if there were >50 spot-forming units (SPU)/50,000 cells observed for NY-ESO-1 peptides and a ≥2-fold increase in SPU compared with a negative control. The induction of an anti-NYESO-1 CD4 or CD8 positive T-cell response was deﬁned as de novo positive or ≥2-fold rise in the number of SPU after the ﬁrst dose. A fluorescence-activated cell sorting (FACS)-based intracellular cytokine staining assay for interferon gamma or tumor necrosis factor alpha after stimulation with NY-ESO-1 peptide was also used and staining ≥2-fold above the baseline value was considered positive for T-cell responses. The number of participants that were anti-NY-ESO-1 T cell positive after induction with treatment is presented.
Time Frame: Up to approximately 24 months
Population: The analysis population included all participants who received ≥1 dose of any of the CMB305 components (LV305, G305) or atezolizumab and had data available for induction after treatment T cell analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 26 | 20
Participants | 14 | 3
Statistical Analysis 1: Comparison: CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab vs Atezolizumab; Test type: Other; p = 0.0127, exact Pearson chi-square test

14. Other Pre Specified Outcome: Overall Response Rate (ORR) Per Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was determined in all participants and was defined as the percentage of participants who had a confirmed Complete Response (CR: Disappearance of all lesions in 2 consecutive observations ≥4 weeks apart) or a Partial Response (PR: ≥30% decrease in tumor burden compared with baseline in 2 observations ≥4 weeks apart) per RECIST 1.1 modified to use irRC confirmation and unidimensional tumor measurements as assessed by BICR. Participants with missing data were considered non-responders. The percentage of participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 36.1 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
Number analyzed (Participants) | 45 | 44
Percentage of participants | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 8.0]

ADVERSE EVENTS:
Time Frame: Up to approximately 36.1 months
Description: Populations: All participants who received ≥1 dose of study treatment for AEs; all randomized participants for all-cause mortality. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 31/45 | 27/44
Serious Adverse Events (participants affected / at risk) | 17/45 | 9/43
Other Adverse Events (participants affected / at risk) | 42/45 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab (N=45) | Atezolizumab (N=43)
Acute left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMB305 (Sequentially Administered LV305 and G305)+Atezolizumab (N=45) | Atezolizumab (N=43)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 6 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (10) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 12 (15) | 7 (11)
Nausea (Gastrointestinal disorders) | 12 (15) | 11 (12)
Vomiting (Gastrointestinal disorders) | 5 (7) | 7 (7)
Chest pain (General disorders) | 4 (4) | 2 (2)
Chills (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 18 (31) | 10 (11)
Influenza like illness (General disorders) | 3 (4) | 3 (4)
Injection site pain (General disorders) | 5 (5) | 0 (0)
Injection site reaction (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 6 (7)
Activated partial thromboplastin time prolonged (Investigations) | 4 (10) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (5) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 4 (9) | 4 (5)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4) | 5 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (6) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (9) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (8)
Headache (Nervous system disorders) | 6 (7) | 7 (7)
Neuralgia (Nervous system disorders) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 5 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Manuscripts reporting the results of this clinical trial, abstracts, press releases, and other media presentations must be provided to the Sponsor for review and comment 30 days prior to submission for publication and may be delayed for up to an additional 30 days in order to ensure that confidential and proprietary data, and intellectual property rights, are protected. Co-authorship of publications will be discussed and mutually agreed upon before submission of a manuscript to a publisher.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT02609984/SAP_000.pdf
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT02609984/Prot_001.pdf